CLINICAL TRIAL: NCT01520311
Title: Post-market Study to Evaluate Post-implant Patency Rates of the eSVS Mesh in the Treatment of Saphenous Vein Graphs During Coronary Artery Bypass Grafting Versus Saphenous Vein Grafts Without the eSVS Mesh Via Coronary Angiography and Duplex Ultra-Sonography Results
Brief Title: The eSVS® Mesh Post-Marketing Trial
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Company closed
Sponsor: Kips Bay Medical, Inc. (Industry)
Collaborators: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO-11015.000 or 297/11 v2.0
Record Dates: First submitted 2012-01-03; First posted 2012-01-27 (Estimated); Last update posted 2016-06-29 (Estimated); Status verified 2016-06

CONDITIONS: Coronary Artery Disease; Myocardial Ischemia; Coronary Disease; Heart Diseases; Cardiovascular Diseases; Arteriosclerosis; Arterial Occlusive Diseases; Vascular Diseases
Keywords: Coronary Artery Disease; Myocardial Ischemia; Coronary Disease; Heart Diseases; Cardiovascular Diseases; Arteriosclerosis; Arterial Occlusive Diseases; Vascular Diseases; CABG; SVG; eSVS Mesh; Bypass Grafting
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia; Coronary Disease; Heart Diseases; Cardiovascular Diseases; Arteriosclerosis; Arterial Occlusive Diseases; Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SVG + eSVS Mesh vs Control SVG (Other): Either the Circumflex Coronary Artery or the Right Coronary Artery will receive the mesh supported vein graft and the native saphenous vein as second and control graft.
  Interventions: Device: eSVS Mesh

INTERVENTIONS:
Device: eSVS Mesh — Patients with multi-vessel coronary artery disease who require SVG CABG of the Right Coronary Artery and the Circumflex Artery due to atherosclerotic Coronary Artery Disease will serve as their own control. They will be randomized to either an SVG+eSVS Mesh to the RCA and an SVG to the Cx or an SVG to the RCA and an SVG+eSVS Mesh to the Cx.
  Other Names: eMesh; external saphenous vein support mesh

SUMMARY:
The purpose of this study is to evaluate patency rates of the eSVS Mesh Saphenous Vein Graph (SVG) and control SVG at six and twenty-four months via coronary angiography and analyses of Duplex Sonography Results and coronary angiography and major cardiovascular or cerebrovascular event (MACCE)-Rate as well as analysis of preoperative great saphenous vein (GSV) duplex sonography and intra-operative GSV harvesting findings and procedure.

DETAILED DESCRIPTION:
This Study will enroll up to 100 patients total. Patients will be enrolled upon meeting certain inclusion criteria, including GSV duplex-sonography results and consent. They will be enrolled based on their clinically indicated requirement for coronary artery bypass grafting with use of their saphenous vein graft. The study will be prospective, randomized repeated measure controlled trial based on the patient's ability to receive both control and eSVS Mesh treatment. Graft patency, MACCE at 6 and 24 months after meshed and non meshed GSV graft implantation will be measured and the findings and qualification of GSV in preoperative duplex sonography will be compared with intraoperative findings while GSV harvesting in order to evaluate the safety of the eSVS mesh and the role of preoperative GSV duplex sonography.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring SVG CABG of the Right Coronary Artery (RCA) AND the Circumflex Artery (Cx) Systems due to atherosclerotic coronary artery disease in both of the two vessels with equal to or greater than 75% stenosis at a single site or multiple stenosis of less than 75%
* Patient with approximately sized and accessible target coronary arteries, with a minimal diameter of 1.5mm and a lack of severe calcification at the anastomotic site
* On-pump, off-pump and beating heart (beating heart with cardiopulmonary bypass) CABG.
* SVG's (eSVS Mesh treated AND non-meshed control vein graft) complying with the size requirements as outlined in the eSVS Mesh "Instructions for Use"
* CABG operational procedure must allow an eSVS Mesh implant procedure as to the eSVS Mesh Instructions for Use
* Patients equal to or greater than 21 years of age
* German language (mother tongue or fully comprehensive patients)
* Any other language with appropriate translation (fully comprehensive patients)
* The patient's accordance to CABG confirmed by a signed standardized internal informed consent for CABG
* Patient able to give their informed written consent

Exclusion Criteria:

* Patients not able to give their informed written consent
* No appropriate target coronary vessel (impaired accessibility, less than 1.5mm diameter, severe calcification)
* SVG's (eSVS Mesh treated AND non-meshed control venous graft) NOT complying with the size requirements as outlined in the eSVS Mesh Instructions for Use
* CABG operational procedure, that DO NOT ALLOW an eSVS Mesh implant procedure as to the eSVS Mesh Instructions for Use
* Concomitant non-CABG cardiac procedure(s)
* Prior cardiac surgery
* Concomitant disease likely to limit life expectancy to less than 2 years
* inability to tolerate or comply with normal post-surgical drug regimen (antiplatelet plus statin)
* Inability to comply with required follow-ups, including angiography imaging methods (allergy to contrast medium, renal insufficiency with creatnine level greater than 150 mmol/l)
* Patients with a known or suspected infection in the field of operation
* Patient is pregnant or intends to become pregnant within 24 months
* Non-pregnant Patient of childbearing potential, who is not prepared for contraception during the study-period
* Concurrent participation in another interventional trial (excluding observational/survey studies)
* Foreign language (no entire comprehension of the patient information and informed study consent guaranteed)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2012-01; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Patency and number of stenosis and their degree in eSVS Mesh SVG versus Control SVG | 24 Months
  Severest degree of graft stenosis (in %; range 0-100) of eSVS Mesh Treated and Non-Meshed control saphenous vein grafts (SVG) assessed by angiography 24 months following CABG.

SECONDARY OUTCOMES:
Incidence of MACCE | 30 Days, 6, 12, and 24 Months
  Incidence of postoperative major adverse cardiac or cerebral events (MACCE): postoperative cerebral stroke, myocardial infarction, (Q wave and non-Q wave), post-implant coronary revascularization (Re-CABG or percutaneous coronary intervention (PCI)) and overall mortality after CABG.
Evaluation and comparison of vein characteristics of SVGs pre-operatively using duplex-sonography versus intraoperatively by standard vein harvest | Baseline
  Pre-operative duplex-sonographic evaluation of the in situ saphenous vein graft charicteristics compared to intra-operative venous harvesting records.

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Reuthebuch, PD Dr. med, Principal Investigator — University Hospital Basel, Clinic for Cardiac Surgery; Devdas Inderbitzin, MD, Study Chair — University Hospital Basel, Clinic for Cardiac Surgery
Locations (1):
- University Hospital, Basel, Switzerland